CLINICAL TRIAL: NCT06885866
Title: Emotion Focused Internet Delivered Treatment for Adults with Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Hugo Hesser, Professor, Linkoeping University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBL-2021-00215
Record Dates: First submitted 2025-02-21; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Eating Disorders
Keywords: Eating disorder treatment; Emotion regulation treatment; Internet treatment
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: A single-case experimental randomized AB-design. Baseline length (i.e., phase A) and start of the B-phase is randomized for each participant. Both phases consist of active treatment, with the purpose of investigating if the interventions added in phase B could enhance treatment results additionally beyond the interventions given during the baseline period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Emotion regulation treatment (Experimental)
  Interventions: Behavioral: Emotion regulation treatment

INTERVENTIONS:
Behavioral: Emotion regulation treatment — Emotion regulation intervention in two phases. Phase A focus on establishing normalised eating patterns, and in phase B the emotion regulation interventions are added. Participants will get access to treatment modules every third day over a time period of 8.5 weeks, each module consist of psychopedagogical material, excercises and home work.

SUMMARY:
The goal of this clinical trial is to develop and test a new internet delivered treatment for adult patients with eating disorders, focused on developing normalized eating patterns and emotion regulation skills. The main focus is to investigate the additional effect of emotion regulation interventions, beyond the effect of other central tratment components normally included in evidence based eating disorder treatment.

The internet delivered treatment is divided into two phases, phase A and phase B. Phase A focus on establishing normalised eating patterns, and in phase B the emotion regulation interventions are added. Participants will get access to treatment modules every third day over a time period of 8.5 weeks, each module consist of psychopedagogical material, excercises and home work.

Data will be collected via the online research platform every third day during the treatment. Data is also collected at more comprehensive assessment points pre-treatment, post-treatment, and follow up 3 months after end of treatment.

DETAILED DESCRIPTION:
This study uses an experimental single-case design, specifically a randomized replicated AB design.

The baseline lenght (i.e., phase A) is randomized for each participant. There is six possible assignments, as the randomization is restricted to give all participants minimum 8 and maximum 12 treatment modules in each phase, with minimum 9 and maximum 14 baseline assessment points.

ELIGIBILITY:
Inclusion Criteria:

* DSM5 eating disorder
* Minimum 18 years old
* Ongoing contact with a psychiatric clinic in sweden

Exclusion Criteria:

* Body mass index below 18,5
* Somatic instability due to eating disorder severeness
* High risk of suicide or severe self-harm
* Ongoing addiction or substance abuse
* Ongoing psychological treatment or psychotherapy
* New or changed mediciation for psychiatric disorders in the past 2 months
* Planned or ongoing pregnancy or recently gave birth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale, 36 items | At pre-treatment assessment one week before treatment start; at post-treatment assessment at day 63 counted from treatment start; and at follow-up assessment at day 153 counted from treatment start.
  Assessment of emotion regulation difficulties. 36 items scored 1-5, higher scores indicate more difficulties. Total score range from 36-180.
Difficulties in Emotion Regulation Scale, 16 items | Counted from treatment start: at day 1, 4, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60
  Assessment of emotion regulation difficulties, short version. 16 items scored 1-5. Higher scores indicates more difficulties. Total score range from 16-80.
The Positive and Negative Affect Schedule, short form | Counted from treatment start: at day 1, 4, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60
  Assessment of affect levels. In this study, only the subscale measuring negative affect is used. 5 items scored 1-5. Higher scores indicate higher levels of negative affect. Total score range from 5-25.

SECONDARY OUTCOMES:
Eating Disorder Examination Questionnaire 6.0 | At pre-treatment assessment one week before treatment start; at post-treatment assessment at day 63 counted from treatment start; and at follow-up assessment at day 153 counted from treatment start.
  Assessment of eating disorder symptoms. 28 items scored 0-6. Higher scores represent more eating disorder pathology. Scores are summerized and scaled, giving a total score ranging from 0-6.
Eating Disorder Symptom List | Counted from treatment start: at day 1, 4, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60
  Assessment of eating disorder symptoms. 8 items scored 0-3, with higher scores indicating more frequent eating disorder symptoms. Total score range from 0-24.
Clinical Impairment Assessment | At pre-treatment assessment one week before treatment start; at post-treatment assessment at day 63 counted from treatment start; and at follow-up assessment at day 153 counted from treatment start.
  Assessment of eating disorder related psychosocial impairment. 16 items scored 0-3. Higher scores indicate higher impairment. Total score range from 0-48.
Clinical Impairment Assessment, subscale social | Counted from treatment start: at day 1, 4, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60
  Assessment of eating disorder related psychosocial impairment, subscale focusing on social impariment.
  5 items scored 0-3. Higher scores indicate higher impairment. Total score range from 0-15.
Normalized eating pattern | Counted from treatment start: at day 1, 4, 9, 12, 15, 18, 21, 24, 27, 30, 33, 36, 39, 42, 45, 48, 51, 54, 57, 60
  Self-assessment of eating patterns, developed by the authors for use in the present study. The self-assessment includes 2 questions:
  1. How many of the previous three days have you eaten regular meals approximately 6 times per day?
  2. How many of the previous three days have you eaten normal sized portions at all or almost all meals?
  Items are scored 0-3. Higher scores indicare more normalized meal habits. Lower scores indicate disordered eating. Total score range from 0-6.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Hesser, PhD, Principal Investigator — Örebro University, Linköping University
Locations (1):
- Linköping University, Linköping, Östergötland County, Sweden

IPD SHARING:
Plan to Share IPD: No
The data set analyzed during the present study is not publicly available, as it contains information that could compromise research participant privacy/consent. However, it could be made available on request to the corresponding author if granted by Swedish Ethical Review Authority.